CLINICAL TRIAL: NCT05633043
Title: Validation of the Cannabis Abuse Screening Test in General Practice(GP-CAST)
Acronym: GP-CAST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 LAPORTE
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-10

CONDITIONS: Cannabis; Addictive Behavior; General Practice; Primary Care; Substance-Related Disorders; Questionnaires
MeSH Terms: conditions — Marijuana Abuse; Behavior, Addictive; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 16-18 year, CAST binary version: Enrollment estimates are based on COSMIN recommendations (https://www.cosmin.nl/) (3). To achieve psychometric validity of the CAST, 110 patients should be included, 50 of whom would be retested. It is proposed to include 110 patients for each of the 3 age categories under study (16-18 years, 18-25 years and 25-45 years) and for each of the 2 scales tested, i.e. a total of 110*3 (age classes)*2 versions of the CAST = 660 patients. In each age category and for each scale: 50 patients (among the 110) will have to complete the Retest phase, i.e. 50*3*2=300 patients (among the 660).
  Five inclusion centers (DMG) will participate in the study, which makes 132 patients per investigating center (66 patients for each scale, i.e. 22 patients for each scale and each age category in each DMG). The GPs will have to include 13.2 patients, during the 12 months of the study.
- 16-18 year, CAST Likert version: Enrollment estimates are based on COSMIN recommendations (https://www.cosmin.nl/) (3). To achieve psychometric validity of the CAST, 110 patients should be included, 50 of whom would be retested. It is proposed to include 110 patients for each of the 3 age categories under study (16-18 years, 18-25 years and 25-45 years) and for each of the 2 scales tested, i.e. a total of 110*3 (age classes)*2 versions of the CAST = 660 patients. In each age category and for each scale: 50 patients (among the 110) will have to complete the Retest phase, i.e. 50*3*2=300 patients (among the 660).
  Five inclusion centers (DMG) will participate in the study, which makes 132 patients per investigating center (66 patients for each scale, i.e. 22 patients for each scale and each age category in each DMG). The GPs will have to include 13.2 patients, during the 12 months of the study.
- 18-25 year, CAST binary version: Enrollment estimates are based on COSMIN recommendations (https://www.cosmin.nl/) (3). To achieve psychometric validity of the CAST, 110 patients should be included, 50 of whom would be retested. It is proposed to include 110 patients for each of the 3 age categories under study (16-18 years, 18-25 years and 25-45 years) and for each of the 2 scales tested, i.e. a total of 110*3 (age classes)*2 versions of the CAST = 660 patients. In each age category and for each scale: 50 patients (among the 110) will have to complete the Retest phase, i.e. 50*3*2=300 patients (among the 660).
  Five inclusion centers (DMG) will participate in the study, which makes 132 patients per investigating center (66 patients for each scale, i.e. 22 patients for each scale and each age category in each DMG). The GPs will have to include 13.2 patients, during the 12 months of the study.
- 18-25 year, CAST Likert version: Enrollment estimates are based on COSMIN recommendations (https://www.cosmin.nl/) (3). To achieve psychometric validity of the CAST, 110 patients should be included, 50 of whom would be retested. It is proposed to include 110 patients for each of the 3 age categories under study (16-18 years, 18-25 years and 25-45 years) and for each of the 2 scales tested, i.e. a total of 110*3 (age classes)*2 versions of the CAST = 660 patients. In each age category and for each scale: 50 patients (among the 110) will have to complete the Retest phase, i.e. 50*3*2=300 patients (among the 660).
  Five inclusion centers (DMG) will participate in the study, which makes 132 patients per investigating center (66 patients for each scale, i.e. 22 patients for each scale and each age category in each DMG). The GPs will have to include 13.2 patients, during the 12 months of the study.
- 25-45 year, CAST binary version: Enrollment estimates are based on COSMIN recommendations (https://www.cosmin.nl/) (3). To achieve psychometric validity of the CAST, 110 patients should be included, 50 of whom would be retested. It is proposed to include 110 patients for each of the 3 age categories under study (16-18 years, 18-25 years and 25-45 years) and for each of the 2 scales tested, i.e. a total of 110*3 (age classes)*2 versions of the CAST = 660 patients. In each age category and for each scale: 50 patients (among the 110) will have to complete the Retest phase, i.e. 50*3*2=300 patients (among the 660).
  Five inclusion centers (DMG) will participate in the study, which makes 132 patients per investigating center (66 patients for each scale, i.e. 22 patients for each scale and each age category in each DMG). The GPs will have to include 13.2 patients, during the 12 months of the study.
- 25-45 year, CAST Likert version: Enrollment estimates are based on COSMIN recommendations (https://www.cosmin.nl/) (3). To achieve psychometric validity of the CAST, 110 patients should be included, 50 of whom would be retested. It is proposed to include 110 patients for each of the 3 age categories under study (16-18 years, 18-25 years and 25-45 years) and for each of the 2 scales tested, i.e. a total of 110*3 (age classes)*2 versions of the CAST = 660 patients. In each age category and for each scale: 50 patients (among the 110) will have to complete the Retest phase, i.e. 50*3*2=300 patients (among the 660).
  Five inclusion centers (DMG) will participate in the study, which makes 132 patients per investigating center (66 patients for each scale, i.e. 22 patients for each scale and each age category in each DMG). The GPs will have to include 13.2 patients, during the 12 months of the study.

SUMMARY:
In France, consumption levels of alcohol, tobacco and cannabis remain high despite changes in regulations aimed at limiting access to these products and repeated prevention campaigns. The various Presidential Plans for the treatment and prevention of addictions for 2007-2011 and 2018-2022 show the concern of the public authorities on the issue of multiple consumption, encouraging general practitioners to identify and research this issue.

In order to better identify and evaluate high-risk cannabis use, the French Observatory for Drugs and Drug Addiction has developed a detection tool: The Cannabis Abuse Screening Test (CAST). Although recommended in France, this questionnaire has never been tested in real primary care conditions, directly with patients consulting general medicine.

The main objective of this study is the validation of a scale for the identification of problematic cannabis use, CAST, with a response modality according to a Likert scale (rated from 0 to 4 : 0 "never", 1 "rarely", 2 "occasionally", 3 "quite often", 4 "very often") or a binary response modality (response by 1 "Yes" or 0 "No") in patients who have used cannabis in the past 12 months, followed in general practice and in 3 age categories (15-18 years, 18-25 years and 25-45 years). The secondary objective is to analyze the polydrug use of alcohol and tobacco, and then the relationship between them and the level of cannabis use.

This validation study of diagnostic scales in real-life situations with general medicine patients allows us to focus on the human and social sciences and public health. Although it has now been established that there is a synergy between several addictive substances with respect to cancer risks, few studies have focused on the early identification of misuse or polydrug use. However, it has been shown that general practitioners (GPs) are effective and relevant players in these fields. Because of their holistic vision of the patient, GPs are in the best position to identify consumers at risk of complications without blaming, dramatizing or trivializing. It is therefore necessary to provide GPs with early detection tools to promote contact between these patients and the healthcare system.

DETAILED DESCRIPTION:
Cannabis is the most widely used illicit substance in France. In order to identify and assess problematic use, the OFDT has developed the Cannabis Abuse Screening Test or CAST.

The French National Authority for Health recommends a tool for early identification and brief intervention for alcohol, cannabis and tobacco use in adults. It includes the CAST questionnaire with YES or NO answers to the questions, but it has not been validated in primary care in this modality (only in a Likert format).

General practitioners therefore do not have a validated tool to screen patients with cannabis use disorder. A quick and efficient tool would allow to optimize the screening practices in general practice by adapting the thresholds of results by sex and age groups.

Primary objective and primary outcome Validation of a Cannabis Abuse Screening Test (CAST) risky cannabis use identification scale with a Likert scale response modality (rated from 0 to 4: 0 "never," 1 "rarely," 2 "occasionally," 3 "quite often," 4 "very often") or a binary response modality (response by 1 "YES" or 0 "NO"), in patients who had used cannabis in the past 12 months, followed up in general practice and among 3 age categories (16-18 years, 18-25 years, 25-45 years).

Secondary objectives and outcome measures

1. To compare the psychometric properties of the CAST according to its 2 response modalities, with respect to their ability to identify early on users with a cannabis use disorder.
2. To determine consumption patterns by age group and their possible links with problematic cannabis use based on the time frame of first use.
3. To analyze the polyconsumption of alcohol, tobacco, e-cigarettes and/or other drugs, and the links between them and cannabis use.
4. To describe patient profiles at risk of cannabis misuse through socio-demographic data, medical data and polyuse.

Schema of the study The objective of this study is to test the CAST questionnaire according to its 2 response modalities, complete and binary. To do this, we will constitute 2 groups of patients: the first will fill in the Cast in binary version (1 "Yes" or 0 "No") and the second will fill in the Likert version. In each of the 2 groups, the 2 versions of the CAST questionnaire will be filled in according to the same procedure: the questionnaire will be filled in by the patient, without any intervention by the physician, at the time of inclusion in general medicine. A questionnaire will be completed 15 days later by the patient at home and returned by mail in a stamped envelope.

Methodology

The following psychometric properties of the CAST scale, in its full and binary versions, will be explored by age categories (16-18 years, 18-25 years, 25-45 years):

* The measure of questionnaire acceptability;
* The reliability (or precision) of the instrument will be assessed according to two criteria: internal consistency and test-retest reproducibility;
* Internal structural validity will explore the consistency of the internal layout of the scale. A factorial analysis approach will complete these analyses;
* The indicators described above (Cronbach, Kappa, correlation coefficient and optimal thresholds) will be systematically compared between the two versions of the CAST scale under study.

Enrollment The size estimate is based on COSMIN recommendations (https://www.cosmin.nl/) (3). To achieve psychometric validity of the CAST, 110 patients should be included, 50 of whom would be retested. It is proposed to include 110 patients for each of the 3 age categories under study (16-18 years, 18-25 years and 25-45 years) and for each of the 2 scales tested, i.e. a total of 110*3 (age classes)*2 versions of the CAST = 660 patients. In each age category and for each scale: 50 patients (among the 110) will have to complete the Retest phase, i.e. 50*3*2=300 patients (among the 660).

Five inclusion centers (DMG) will participate in the study, which makes 132 patients per investigating center (66 patients for each scale, i.e. 22 patients for each scale and each age category in each DMG). The GPs will have to include 13.2 patients, during the 12 months of the study.

Inclusion criteria Patients aged 16 to 45 years, Patients with cannabis use in the past 12 months, Patients followed in general medicine, Patients able to give free and informed consent to participate in the research, Patients affiliated to the French Social Security.

Non-inclusion criteria Patients who started using cannabis less than 12 months ago, Cessation of cannabis use on the day of the test phase (no Retest phase possible), Patients in the process of withdrawal (risk of being withdrawn during the Retest phase), Patients undergoing treatment in an addiction care and prevention center (CSAPA), Patients with decompensated psychosis, Patients unable to complete the questionnaire on their own or with difficulties in understanding the French language, Patients refusing to participate in the research.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 16 to 45 years, Patients with cannabis use in the last 12 months, Patients followed in general medicine, Patients able to give free and informed consent to participate in the research, Patients affiliated to the French Social Security.

Exclusion Criteria:

Patients who started using cannabis less than 12 months ago, Stop using cannabis on the day of the test phase (no Retest phase possible), Patients in the process of withdrawal (risk of being withdrawn during the Retest phase), Patients undergoing treatment in an addiction care and prevention center (CSAPA), Patients with decompensated psychosis, Patients unable to complete the questionnaire on their own or with difficulties in understanding the French language, Patients refusing to participate in the research.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Test phase: Patients will be recruited from the active file of general practitioners participating in the study and according to the specified inclusion criteria. An information letter outlining the objectives of the study will be given to the patients and the physician will inform them that the data will be anonymized and will remain strictly confidential. The patient will be informed that his or her decision to participate in the study or not will not affect his or her treatment. The patient will also be informed of his or her right to withdraw from the study at any time without justification and without consequence on his or her care.
  Retest phase: The patient must return the completed CAST scale (in the same format as the one submitted during the inclusion consultation) within a maximum of 2 to 4 weeks by mail to the coordinating center in a pre-stamped envelope provided. He/she will receive financial compensation upon receipt of the Retest questionnaire.
Sampling Method: Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Validation of a Cannabis Abuse Screening Test (CAST) in general practice | 12 months
  Validation of a Cannabis Abuse Screening Test (CAST) with a Likert scale response modality (rated from 0 to 4: 0 "never," 1 "rarely," 2 "occasionally," 3 "quite often," 4 "very often") or a binary response modality (response by 1 "YES" or 0 "NO"), in patients who had used cannabis in the past 12 months, followed up in general practice and among 3 age categories (16-18 years, 18-25 years, 25-45 years).

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Département de Médecine Générale de Clermont-Ferrand, Clermont-Ferrand
  - Département de Médecine Générale de Grenoble, Grenoble
  - Département Universitaire de Médecine Générale, Lyon, Lyon
  - Département de Médecine Générale de Saint-Etienne, Saint-Etienne
  - Département Universitaire de Médecine Générale, Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No